CLINICAL TRIAL: NCT00859417
Title: PERIGEE :Randomized Study Evaluating the Effectiveness of the Use of Prosthesis With Trans-obturator Way for the Correction of Anterior Prolapse.
Brief Title: Study Evaluating the Effectiveness of the Use of Prosthesis With Trans-Obturator Way for the Correction of Anterior Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007.485/28
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2013-11

CONDITIONS: Anterior Prolapse
Keywords: correction of anterior prolapse; prosthetic trans-obturator way kit; randomized study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Traditional surgical method without prosthesis
  Interventions: Procedure: Traditional surgery
- 2 (Experimental): Surgical method with Perigee prosthesis
  Interventions: Device: Perigee® prosthesis

INTERVENTIONS:
Procedure: Traditional surgery — Traditional surgical method without prosthesis (correction of the anterior prolapse through vaginal tract with the use of autologous tissue).
  Arms: 1
Device: Perigee® prosthesis — Surgical method with Perigee® prosthesis
  Arms: 2

SUMMARY:
The classical surgical treatment of an anterior prolapse is the use of autologous tissue. In front of the high rate of recurrences with this technique, the use of synthetic prosthesis made their appearance. But the drawback of the use of prosthesis is their tolerability. The system Perigee®, a prosthetic kit by trans-obturator way, was designed to obtain high efficiency in the correction of the prolapse while reducing the risk of complications. The lack of prospective and randomized studies makes difficult to assess the interest. The investigators, therefore, have put in place a randomized prospective study seeking the evaluation of the system Perigee® compared to the conventional surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Genital anterior prolapse requiring surgical correction and with stage III or IV in the classification of Pelvic Organ Prolapse - Quantification or POP-Q
* Ability to understand the information and to sign a consent form
* Patients wishing an intervention because of the inconvenience caused by the prolapse.

Exclusion Criteria:

* Prolapse stage <III in the classification POP-Q, and prolapse without functional inconvenience
* Progressive or latent infection, or signs of tissue necrosis in the clinical examination
* Troubles resulting in an unacceptable risk of post-surgery complications investigated at the interview with the patient (disorders of blood clotting, immune system disorders, progressive diseases….)
* Mobility of the lower limbs reduced (not permitting the positioning for the surgery)
* Pregnancy or any desire of pregnancy during the study, within two years
* Pelvic surgery in the last 6 months
* Patients who have had radiotherapy of the pelvic area in an irrespective time
* A history of pelvic cancer
* Known hypersensitivity to any component of the prosthesis (polypropylene)
* Uncontrolled diabetes (HbA1c> 8%)
* Treatment modifying the immune response (immuno-modulators), current or stopped for less than one month
* Inability to understand the information and to sign a consent
* A person not subject to social security, deprived of freedom, or under legal guardian

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Correction of prolapse, which is defined by a stage < II on the classification POP-Q, one year after surgery | 12 months

SECONDARY OUTCOMES:
Correction of prolapse 2 years after surgery | 24 months
Changes in quality of life, occurrence of complications during surgery, evolution of sexuality, onset or worsening of urinary incontinence | at 3,12, 24 months
Pain after surgery | 24 months
Duration of intervention | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MELLIER Georges, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital femme Mère Enfant, Bron, France

REFERENCES:
- [Result] Lamblin G, Van-Nieuwenhuyse A, Chabert P, Lebail-Carval K, Moret S, Mellier G. A randomized controlled trial comparing anatomical and functional outcome between vaginal colposuspension and transvaginal mesh. Int Urogynecol J. 2014 Jul;25(7):961-70. doi: 10.1007/s00192-014-2344-7. Epub 2014 Feb 27. PMID 24573358